CLINICAL TRIAL: NCT03167359
Title: A Pilot Study of Hypofractionated Simultaneous Integrated Boost Radiotherapy in Stage 0, I and III Breast Cancer Patients
Brief Title: Hypofractionated Radiotherapy in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Mylin Torres, MD, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00047240
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Cancer, Breast; Inflammation
Keywords: Psychiatry; Radiation Therapy
MeSH Terms: conditions — Breast Neoplasms; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Participants with Stage 0-III breast cancer (Experimental): Women with Stage 0-III breast cancer, treated with breast conserving surgery or mastectomy and clear margins, will receive 15 doses of radiation over three weeks.
  Interventions: Radiation: Hypofractionated Simultaneous Integrated Boost Radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated Simultaneous Integrated Boost Radiotherapy — Participants will receive radiotherapy treatments to the whole breast or chest wall to a dose of 2.66 Gy per day x 15 fractions simultaneously with a boost treatment. The boost treatment will be given on the same days as the whole breast treatment. The lumpectomy cavity + scar (in lumpectomy patients) or chest wall scar (mastectomy patients) will receive 0.54 Gy per day x 15 fractions.

SUMMARY:
As the number of breast cancer (BrCA) survivors has markedly increased, clinicians are now seeking to reduce treatment-related toxicities and inconveniences of treatment, namely the traditional 6 weeks of daily radiation treatment (XRT). Skin thickening, fibrosis, and edema are some of the most common acute and potentially long-term debilitating toxicities of BrCA XRT.

The purpose of this study is to learn if three weeks of daily radiation treatment (RT) to the breast is safe in breast cancer patients who are usually prescribed 6 weeks of daily radiation after breast surgery (e.g. lumpectomy or mastectomy) as standard of care.

DETAILED DESCRIPTION:
As the number of breast cancer (BrCA) survivors has markedly increased, clinicians are now seeking to reduce treatment-related toxicities and inconveniences of treatment, namely the traditional 6 weeks of daily radiation treatment (XRT). Skin thickening, fibrosis, and edema are some of the most common acute and potentially long-term debilitating toxicities of BrCA XRT.

The purpose of this study is to learn if three weeks of daily radiation treatment (RT) to the breast is safe in breast cancer patients who are usually prescribed 6 weeks of daily radiation after breast surgery (e.g. lumpectomy or mastectomy) as standard of care.

Investigators seek to assess the rate of cutaneous toxicity, the rates of lymphedema determined by arm measurements and Grade 3 brachial plexopathy in patients receiving regional nodal irradiation, as well as local control, quality of life, and fatigue levels.

ELIGIBILITY:
Inclusion Criteria:

Participants must have one or more of the following characteristics and be eligible for breast or chest wall with or without regional nodal radiotherapy:

* Prior Chemotherapy for Breast Cancer
* Greater than 25 cm of breast separation (the largest distance on an axial slice of the planning CT simulation scan between the entry and exit points of the radiation beam on the body)
* Non-Caucasian Race
* Less than or equal to 50 years of age
* Requiring regional nodal irradiation without evidence of N3 disease

Exclusion Criteria:

* Males will be excluded
* Women who are pregnant or nursing a child may not take part in this study

Max Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mylin Torres, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Stage 0-III Breast Cancer
Started | 74
Completed | 72
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 39
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Per Cutaneous Toxicity Grade (0, 1, 2, 3, 4)
Description: Cutaneous toxicity rate will be assessed by the National Cancer Institute - Common Toxicity Criteria (NCI-CTC) v.3 grading scale. THe NCI CTCAE grades go from 0 to 4. Grade 0: none. Grade 1: Mild or localized; topical intervention indicated. Grade 2: Intense or widespread; intermittent; skin changes from scratching (e.g., edema, papulation, excoriations, lichenification, oozing/crusts); limiting instrumental ADLs. Grade 3-4: Severe or life-threatening. The higher the grade, the worse the outcome.
Time Frame: Duration of Study (Up to 18 months)
Population: Data is missing on one participant who completed the study. Another patient developed a contralateral breast cancer during the study and another patient was lost to follow up. These latter two patients did not complete the 1 year post radiation assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 71
Participants
  Grade 0 | 60
  Grade 1 | 11
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

2. Primary Outcome: Number of Participants With 20% or Greater Increase in Arm Lymphedema Compared to Baseline
Description: Number of Participants with 20% or greater increase in arm lymphedema (compared to baseline arm measurements) will be assessed among breast cancer patients receiving regional nodal irradiation.
Time Frame: Duration of Study (Up to 18 months)
Population: 30 patients received regional nodal irradiation, and per protocol, this subcohort of patients were assessed for lymphedema and brachial plexopathy. Patients who did not receive regional nodal irradiation did not undergo assessments for brachial plexopathy or lymphedema.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 30
Participants | 0

3. Primary Outcome: Number of Participants With Grade 3 Brachial Plexopathy
Description: Number of Participants with Grade 3 Brachial Plexopathy will be assessed among breast cancer patients receiving regional nodal irradiation by RTOG and LENT/SOMA scales Brachial plexopathy range minimum 0 and maximum 4. The higher the score, the worse the outcome
Time Frame: Duration of Study (Up to 18 months)
Population: Per protocol, only patients who received regional nodal irradiation were assessed for brachial plexopathy. 30 enrolled patients received regional nodal irradiation and then were assessed for brachial plexopath.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 30
Participants | 0

4. Secondary Outcome: Change in Cutaneous Toxicity Rate Assessed by Ultrasound Tissue Characterizations (UTC)
Description: Ultrasound tissue characterization (UTC) is driven by knowledge of the physics of ultrasound and its interactions with biological tissue, and has traditionally used signal modelling and analysis to characterize and differentiate between healthy and diseased tissue. Change in mean UTC at last assessment (up to 18 months post XRT) was compared to baseline (pre-XRT) measures.
Time Frame: Baseline, end of Follow Up (Up to 18 months) (up to 18 months)
Population: One patient did not complete her ultrasound measurements of skin toxicity.
Measure: Mean (Standard Deviation); unit: percentage change in skin thickness
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 71
percentage change in skin thickness | -0.91 (0.39262)

5. Secondary Outcome: Change in Tumor Necrosis Factor (TNF) - Alpha Levels
Description: Blood will be analyzed for TNF-alpha (TNF)-alpha levels and correlated to the development of cutaneous toxicity.
Time Frame: Baseline, Post Intervention (Up to 18 Months)
Population: Specimens were not processed due to limited funds
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Soluble TNF Receptor 2 (sTNFR2) Levels
Description: Blood will be analyzed for soluble TNF receptor 2 (sTNFR2) levels and correlated to the development of cutaneous toxicity.
Time Frame: Baseline, Post Intervention (Up to 18 Months)
Population: Specimens were not processed due to limited funds.
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Interleukin (IL)-6 Levels
Description: Blood will be analyzed for interleukin (IL)-6 levels and correlated to the development of cutaneous toxicity.
Time Frame: Baseline, Post Intervention (Up to 18 Months)
Population: Specimens were not processed due to limited funds
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Interleukin 1 Receptor Agonist (IL-1ra) Levels
Description: Blood will be analyzed for IL-1ra levels and correlated to the development of cutaneous toxicity.
Time Frame: Baseline, Post Intervention (Up to 18 Months)
Population: Specimens were not processed due to limited funds
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in C - Reactive Protein (CRP) Levels
Description: Blood will be analyzed for CRP levels and correlated to the development of cutaneous toxicity.
Time Frame: Baseline, Post Intervention (Up to 18 Months)
Population: Specimens were not processed due to limited funds
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Multidimensional Fatigue Inventory (MFI) Score
Description: The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure fatigue. Scores range from 20 to 100.The higher the score, the more fatigued. The higher the maximum change, the greater increase in fatigue a patient feels.
Time Frame: Baseline, end of Follow Up (Up to 18 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 72
score on a scale | -6.33 (12.96)

11. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) Score
Description: The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Scores range from 0 to 21. A score of less than or equal to 5 is associated with good sleep quality. A score greater than 5 is associated with poor sleep quality. The higher the maximum change, the greater increase in sleep disturbances a patient has.
Time Frame: Baseline, End of Follow Up (Up to 18 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 72
score on a scale | -0.75 (2.77)

12. Secondary Outcome: Change in Perceived Stress Scale (PSS) Score
Description: The PSS is a self-reported instrument used to measure the perception of stress. Scores range from 0 to 40. Score of 20 or higher are considered high stress. The higher the maximum change, the greater increase in stress the patient feels.
Time Frame: Baseline, End of Follow Up (Up to 18 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 72
score on a scale | -2.92 (6.99)

13. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form Score
Description: The PROMIS Fatigue questionnaire is a self-report tool used to evaluate frequency, duration, and intensity of fatigue over the past seven days. Scores range from 7 to 35. The higher the score, the more fatigue.
Time Frame: Baseline, End of Follow Up (Up to 18 months)
Population: Patient were asked to complete this instrument only after an amendment was made to the protocol. Therefore, the last 23 patients enrolled completed this survey due to the fact that it was added to the protocol in after the majority of patients had been enrolled on the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 23
score on a scale | -2.57 (6.82)

14. Secondary Outcome: Change in an Inventory of Depressive Symptomatology-Self Reported (IDS-SR) Score
Description: The IDS-SR is a self-reported measure in which participants rate the frequency of depression symptoms within the past seven days. Scores range from 0 to 84, with higher score reflecting greater severity of depressive symptoms.
Time Frame: Baseline, End of Follow Up (Up to 18 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 72
score on a scale | -3.21 (8.81)

15. Secondary Outcome: Change in Short Form-36 (SF-36) Health Survey Score
Description: The SF-36 is a self-reported survey of health status. Scores range from 0 to 100. Lower scores indicate disability. The higher the score, the less disability.
Time Frame: Baseline, End of Follow Up (Up to 18 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 72
score on a scale | 11.07 (15.89)

16. Secondary Outcome: Change in Godin Leisure-Time Exercise Questionnaire (GLTEQ) Score
Description: The GLTEQ is a self-reported questionnaire used to measure usual leisure-time exercise habits during a typical seven day period. The GLTEQ specifically inquires about frequency of mild, moderate, and strenuous physical activity done during a typical 7-day period with exercise of more than 15 min or more per day during the previous week.
  Total score for the Godin leisure-time exercise questionnaire is calculated using this formula.Weekly leisure activity score = (9 × Strenuous) + (5 × Moderate) + (3 × Light).
  The GLTEQ total score can be broken into three categories:
  less than 14 points = sedentary 14 - 23 points is = moderately active 24 points or more = active The score ranges from 0 to 119.
Time Frame: Baseline, End of Follow Up (Up to 18 months)
Population: This instrument was added to the protocol in an amendment and therefore the first two patients who were enrolled did not complete this instrument because they participated prior to approval of that amendment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 70
score on a scale | 5.21 (21.55)

17. Secondary Outcome: Change in Lent Soma Scale Patient Questionnaire Score
Description: The Lent Soma questionnaire is a self-reported measure of pain. Scores range from 0 to 9. The higher the score, the more pain reported.The higher the maximum change, the more increase in breast pain, the patient is perceiving.
Time Frame: Baseline, End of Follow Up (Up to 18 months)
Population: Per protocol, this questionnaire was administered only to patients who received regional nodal irradiation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 30
score on a scale | -1.12 (2.59)

18. Secondary Outcome: Change in Breast Pain Level
Description: Participants will be asked to rate their breast pain level on a study specific scale from 0 to 10 where 0 represents no pain, and 10 represents the most extreme pain. The higher the maximum change, the more increase in breast pain, the patient is perceiving.
Time Frame: Baseline, End of Follow Up (Up to 18 months)
Population: This instrument was added in an amendment to the protocol after a number of patients had already been enrolled. Once approved, patients who were enrolled then completed the instrument at the corresponding timepoints after the amendment was approved.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 57
score on a scale | 0.26 (2.51)

19. Secondary Outcome: Change in Breast Appearance Satisfaction Score
Description: Participants will be asked to rate the look of their breast on a study specific scale from 0 to 10 where 0 represents not happy, and 10 represents very happy. The higher the maximum change, the more increase in happiness with breast appearance the patient is reporting.
Time Frame: Baseline, End of Follow Up (Up to 18 months)
Population: This questionnaire was added in an amendment after the majority of patients were enrolled on study. Once the amendment was approved by Emory IRB, the questionnaire was administered to the remaining 33 patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 33
score on a scale | .30 (2.62)

20. Secondary Outcome: Change in Radiated Breast Appearance Score
Description: Participants will be asked to rate how different the look of their radiated breast is compared to their non-radiated breast on a study specific scale from 0 to 10 where 0 represents no difference, and 10 represents completely different.
Time Frame: Baseline, End of Follow Up (Up to 18 months)
Population: This questionnaire was added as an amendment after the majority of patients had been enrolled and assessed. Once the amendment was Emory IRB approved, the questionnaire was administered to the remaining 31 patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Stage 0-III Breast Cancer
Number analyzed (Participants) | 31
score on a scale | -0.81 (4.02)

ADVERSE EVENTS:
Time Frame: 60 months
Arm/Group | Participants With Stage 0-III Breast Cancer
All-Cause Mortality (participants affected / at risk) | 2/74
Serious Adverse Events (participants affected / at risk) | 3/74
Other Adverse Events (participants affected / at risk) | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Stage 0-III Breast Cancer (N=74)
Recurrance (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT03167359/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03167359/SAP_001.pdf